CLINICAL TRIAL: NCT07214753
Title: ItAlian, Multicenter, Observational, Prospective sTudy to Evaluate the acHievement of Clinical rEmission and immuNomodulation in Severe Eosinophilic Asthma Patients Treated With Benralizumab - the ATHENA Study
Brief Title: A Real-life Observational Study in Severe Eosinophilic Asthma Adult Participant Treated With Benralizumab in Italy
Acronym: ATHENA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00141
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: benralizumab — 30mg s.c. as per SmPC
  Other Names: Fasenra

SUMMARY:
This is an observational, multicenter, prospective study on patients with severe eosinophilic asthma treated with benralizumab aimed at evaluating the achievement of partial and complete clinical remission.

DETAILED DESCRIPTION:
The ATHENA study aims to expand real-world evidence on benralizumab role in clinical practice, specifically evaluating its effectiveness in achieving clinical remission (complete and partial), as defined by SANI. Additionally, given the growing importance of biomarkers in asthma research, this study seeks to further investigate benralizumab immunological effects, potentially contributing to a deeper understanding of asthma pathophysiology and addressing existing knowledge conundrum. Additionally, the study will consolidate long-term safety data.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old) diagnosed with severe uncontrolled eosinophilic asthma.
* Benralizumab has been prescribed according to the approved label and local reimbursement criteria
* Provision of signed Informed Consent Form (ICF) prior to any study-related activities
* Benralizumab has been initiated within 7 days prior to study enrollment or is planned to be initiated within 7 days after enrollment (in the latter case, provided that the decision to prescribe benralizumab is made prior to the decision to enroll the patient in the study).

Exclusion Criteria:

* Benralizumab treatment within the 12 months prior to study enrollment and up to 8 days before enrollment
* Previous participation (in the 12 months before enrollment), current participation or plan to participate within the follow up period to any other clinical trial.
* Contraindication to benralizumab as per current Summary of Product Characteristics (SmPC).
* Pregnant or lactating women.
* patients with any clinical condition that may interfere with the subject's ability to cooperate and comply with the study procedures based on the Investigator's judgement.
* Previous or concomitant use of omalizumab, reslizumab, dupilumab, tezepelumab or mepolizumab without washout period as per clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe eosiniphilic asthma patients treated with benralizumab as per clinical practices
Sampling Method: Non-Probability Sample
Enrollment: 335 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of patients achieving clinical remission, partial and complete, as per SANI Definition | 24 months
  Number and percentage of patient who met the 4 remission criteria (complete or partial) at 12 months and maintained up to 24months

SECONDARY OUTCOMES:
Number and percentage of patients achieving the criteria for clinical remission | 3, 6, 12 and 24 months
  Number and percentage of patient with the criteria for complete or partial remission according to the following criteria: No need to use OCS; Absence of asthma symptoms (ACT score from 20/25 to 25/25); Absence of asthma exacerbations; Stable lung function (FEV1 decline of no more than 100 mL).
Rate of any and SA exacerbations | 3, 6, 12 and 24 months
  annualized exacerbations rate
Mean change in Asthma Control Test (ACT) score | 1, 3, 6, 12 and 24 months vs baseline
  mean (SD) changes (min - max) overtime in ACT score
Mean changes in Asthma Control Questionnaire (ACQ) score | 1, 3, 6, 12 and 24 months vs baseline
  mean (SD) changes (min - max) overtime in ACQ score
Mean change in FEV1 - pre-BD | 3, 6, 12 and 24 vs baseline
  mean (SD) changes in FEV1 (L) overtime
Mean changes in FEV1 - post-BD | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in FEV1 (L) post-BD
Mean changes in FEV1 % predicted - pre-BD | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in FEV1 % predicted pre-BD
Mean changes in FEV1 % predicted - post-BD | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in FEV1 % predicted post-BD
Mean changes in FVC pre-BD | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in FVC (L) pre-BD
Mean changes in FVC post-BD | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in FVC (L) post-BD
Mean changes in pre-BD FEV1/FVC | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in pre-BD FEV1/FVC (ratio)
Mean changes in pre-BD FEF 25-75 | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in pre_BD FEF25-75 (L/sec)
Mean changes in post-BD FEF 25-75 | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in post-BD FEF25-75 (L/sec)
Mean changes in post-BD FEV1/FVC | 3, 6, 12 and 24 months vs baseline
  mean (SD) changes in post-BD FEV1/FVC (ratio)
Change in inhaled maintenance therapy and inhaled corticosteroid (ICS/LABA/LAMA, ICS/LABA) use and dosage | 3, 6, 12 and 24 months
  Change in inhaled maintenance therapy and inhaled corticosteroid (ICS/LABA/LAMA, ICS/LABA) use and dosage after benralizumab treatment
Change in mOCS use and daily dose | 3, 6, 12 and 24 months
  Change in mOCS use and daily dose after benralizumab administartion

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - AZIENDA ULSS 6 EUGANEA_OSPEDALE DI CITTADELLA U.O.C. di Pneumologia, Cittadella, Padova
  - PRESIDIO OSPEDALIERO SANTA MARIA DELLA SPERANZA U.O.C. Medicina Interna, Battipaglia, Salerno
  - OSPEDALE MARIA S.S. DELLO SPLENDORE U.O.S.D. Allergologia Territoriale presidio ospedaliero Giulianova, Giulianova, Teramo
  - AULSS2 MARCA TREVIGIANA OSPEDALE CIVILE DI MONTEBELLUNA U.O.C. di Pneumologia, Montebelluna, Treviso
  - IRCCS MAUGERI TRADATE U.O.di Pneumologia Riabilitativa, Tradate, Varese
  - POLICLINICO DI BARI U.O.C. Malattie dell'Apparato Respiratorio, Bari
  - ASST PAPA GIOVANNI XXIII U.O.C. Pneumologia, Bergamo
  - IRCSS AZIENDA OSPEDALIERO UNIVERSITARIA DI BOLOGNA, POLICLINICO SANT'ORSOLA MALPIGHI U.O. Pneumologia e Terapia intensiva respiratoria, Bologna
  - OSPEDALE BELLARIA U.O.C. Pneumologia, Bologna
  - ASST SPEDALI CIVILI DI BRESCIA S.S.D. Centro Fibrosi Cistica, Brescia
  - AZIENDA OSPEDALIERO UNIVERSITARIA POLICLINICO "G. RODOLICO- SAN MARCO" CATANIA U.O.C Pneumologia, Catania
  - AZIENDA OSPEDALIERO UNIVERSITARIA MATER DOMINI U.O. Pneumologia, Catanzaro
  - AZIENDA OSPEDALIERO UNIVERSITARIA CAREGGI S.O.D. Immuno Allergologia, Florence
  - AZIENDA OSPEDALIERO UNIVERSITARIA POLICLINICO RIUNITI DI FOGGIA S.C. Malattie dell'Apparato Respiratorio, Foggia
  - AZIENDA OSPEDALIERA UNIVERSITARIA POLICLINICO "G.MARTINO" DI MESSINA U.O.S.D. Allergologia ed Immunologia Clinica, Messina
  - ASST SANTI PAOLO E CARLO U.O.C. di Pneumologia, Milan
  - AZIENDA OSPEDALIERO UNIVERSITARIA POLICLINICO DI MODENA S.C. Malattie dell'apparato respiratorio, Modena
  - AZIENDA OSPEDALIERA RILIEVO NAZIONALE COLLI MONALDI U.O.C. Pneumotisiologia Università Federico II, Napoli
  - AZIENDA OSPEDALIERO UNIVERSITARIA FEDERICO II U.O.S.D. Allergologia ed Immunodeficienza, Napoli
  - AZIENDA OSPEDALIERA UNIVERSITA' PADOVA U.O.C Fisiopatologia Respiratoria, Padua
  - AZIENDA OSPEDALIERA UNIVERSITARIA POLICLINICO PAOLO GIACCONE U.O.C. Pneumologia, Palermo
  - FONDAZIONE IRCSS POLICLINICO SAN MATTEO U.O.C. Pneumologia, Pavia
  - AO SAN CAMILLO FORLANINI U.O.S.D. Day Hospital Pneumologico e Interstiziopatie Polmonari, Roma
  - AZIENDA OSPEDALIERO UNIVERSITARIA SANT'ANDREA U.O.C Malattie Apparato Respiratorio, Roma
  - AZIENDA OSPEDALIERO UNIVERSITARIA SASSARI U.O.C. Pneumologia e Interventistica Cliniche San Pietro, Sassari
  - AZIENDA OSPEDALIERO UNIVERSITARIA SENESE U.O.C. Malattie dell'apparato Respiratorio e Trapianto Polmonare, Siena
  - AZIENDA OSPEDALIERA ORDINE MAURIZIANO S.C.D.U. Immunologia e Allergologia, Torino
  - AZIENDA OSPEDALIERA UNIVERSITARIA INTEGRATA-BORGO ROMA U.O. Allergologia e Asma center, Verona